CLINICAL TRIAL: NCT04641429
Title: Neuroplasticity: The Effects of Exercise Training on Cognitive and Affective Functioning of Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Tatia Mei-chun LEE, Chair Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 19-005
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Healthy Ageing
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: In this intervention study, each participant is allocated to either the Qigong or stretching exercise training group in a pseudo-randomized order based on the recruitment orders and their availability.
Masking Description: Blinding the participants to the allocation is impossible due to the nature of intervention. But prior to the first training session, participants have no knowledge on which type of training they are going to receive.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong (Experimental): Participants in the experimental group receive Qigong exercise training.
  Interventions: Behavioral: Qigong exercise
- stretching (Active Comparator): Participants in the control group receive stretching exercise training.
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Qigong exercise — Participants in the experimental group receive 12-week group-based Qigong exercise training.
  Arms: Qigong
Behavioral: Stretching exercise — Participants in the control group receive 12-week group-based stretching exercise training.
  Arms: stretching

SUMMARY:
This study investigates the effects of exercise on older people's cognitive and affective functions, and the possible underlying neurobiological pathways.

DETAILED DESCRIPTION:
Population aging is accelerating. The socioeconomic burden associated with an aging population calls for timely action for promoting brain health. The human brain has the capacity for plastic reorganization through learning and experience. Physical activity could induce plasticity and is important in the prevention of functional decline and increased survival. In this study, the effects of Qigong and stretching exercise on affective and cognitive function among the healthy elderly are investigated. This study is proposed to invite 200 participants (100 in each intervention condition). The investigators acquire data from questionnaires, assessments, neurocognitive tests, magnetic resonance imaging and blood samples at baseline (before the intervention) and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. At least finished primary school;
2. Have normal or corrected-to-normal vision and hearing;
3. Ability to do exercise;
4. Right-hand dominance;
5. Normal cognitive ability as assessed by the Montreal Cognitive Assessment Hong Kong version (HK-MoCA).

Exclusion Criteria:

1. Abmormal anxiety or depression mood as measured by the Hospital Anxiety and Depression Scale;
2. Current diagnosis or history of neurological or psychological conditions, such as substance abuse, psychotic disorders, or affective disorders;
3. Current diagnosis or history of substance/alcohol abuse;
4. Contraindications for MRI scanning (e.g. implanted metal);
5. People who regularly practice any qigong, Tai Chi or similar exercise or meditation within 6 months before study;
6. People who regularly practice moderate to high intensity physical exercise within 6 months before study. The operational definition of 'regular practice' is three times a week or more, at least 30 mins per time for at least 3 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline in cognitive processing speed scores on the Symbol Digit Modalities Test at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of cognitive processing speed scores are measured by the Symbol Digit Modalities Test from baseline to end of intervention at 12 Weeks. Scores on the Symbol Digit Modalities Test range from 0-90, with a higher score indicating better performance.
Mean change from Baseline in sustained attention scores on the Continuous Performance Test at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of sustained attention scores are measured by the Continuous Performance Test from baseline to end of intervention at 12 weeks. The accuracy scores on the Continuous Performance Test range from 0-100%, with a higher score indicating better performance.
Mean change from Baseline in working memory scores on the Digit Span-Backward Test at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of working memory scores are measured by the Digit Span Backward Test from baseline to end of intervention at 12 weeks. Scores on the Digit Span-Backward test range from 2-13, with a higher score indicating better performance.
Mean change from Baseline in language scores on the Rapid Naming Test at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of language scores are measured by the Rapid Naming Test from baseline to end of intervention at 12 weeks. Scores on the Rapid Naming Test range from 0-36, with a higher score indicating better performance.
Mean change from Baseline in trait affect scores on the Chinese Affect Scale at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of trait positive affect and negative affect are measured by the Chinese Affect Scale from baseline to end of intervention at 12 weeks. Positive and negative affect scores on Chinese Affect Scale both range from 10-50, with a higher score indicating higher positive/negative affect.
Mean change from Baseline in affective processing by the Emotion Processing Task at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of affective stimuli processing are measured by the Emotion Processing Task from baseline to end of intervention at 12 weeks.
Mean change from Baseline in blood levels of cortisol at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of blood biomarker levels of cortisol are measured from baseline to end of intervention at 12 weeks.
Mean change from Baseline in blood levels of interleukin-6 at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of blood biomarker levels of interleukin-6 are measured from baseline to end of intervention at 12 weeks.
Mean change from Baseline in blood levels of brain-derived neurotrophic factor at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of blood biomarker levels of brain-derived neurotrophic factor are measured from baseline to end of intervention at 12 weeks.
Mean change from Baseline in telomerase activity at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of blood measurement of telomerase activity are measured from baseline to end of intervention at 12 weeks.
Mean change from Baseline in brain structure by magnetic resonance imaging at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of brain structure are measured by T1-weighted magnetic resonance imaging from baseline to end of intervention at 12 Weeks.
Mean change from Baseline in brain function by functional magnetic resonance imaging at 12 Weeks | from baseline to end of intervention at 12 weeks
  Changes of brain function are measured by functional magnetic resonance imaging from baseline to end of intervention at 12 Weeks.

SECONDARY OUTCOMES:
Mean change from Baseline in perceived stress scores on the Perceived Stress Scale at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of perceived stress scores are measured by the Perceived Stress Scale from baseline to end of intervention at 12 weeks. Scores on the Perceived Stress Scale range from 0-56, with a higher score indicating higher perceived stress.
Mean change from Baseline in insomnia severity scores on the Insomnia Severity Index at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of insomnia severity scores are measured by the Insomnia Severity Index from baseline to end of intervention at 12 weeks. Scores on the Insomnia Severity Index range from 0-28, with a higher score indicating more severe insomnia.
Mean change from Baseline in quality of sleep on the Pittsburg Seep Quality Index at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of quality of sleep scores are measured by the Pittsburg Seep Quality Index from baseline to end of intervention at 12 weeks. Scores on the Pittsburg Seep Quality Index range from 0-21, with a higher score indicating more severe sleeping difficulty.
Mean change from Baseline in depression and anxiety scores on the Hospital Anxiety and Depression Scale at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of depression and anxiety scores are measured by the Hospital Anxiety and Depression Scale from baseline to end of intervention at 12 weeks. Anxiety and Depression scores on the Hospital Anxiety and Depression Scale both range from 0-21, with a higher score indicating more severe anxiety/depression mood.
Mean change from Baseline in perceived loneliness scores on the UCLA Loneliness Scale at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of perceived loneliness scores are measured by the UCLA Loneliness Scale from baseline to end of intervention at 12 weeks. The scores on the UCLA Loneliness Scale range from 20-80, with a higher score indicating greater perceived loneliness.
Mean change from Baseline in quality of life scores on the WHO Quality of Life-BREF scale at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of quality of life scores are measured by the WHO Quality of Life-BREF scale from baseline to end of intervention at 12 weeks. The scores on the WHO Quality of Life-BREF scale range from 26-130, with a higher score indicating higher quality of life.
Mean change from Baseline in emotion reactivity scores on the Emotion Reactivity Scale at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of emotion reactivity scores are measured by the Emotion Reactivity Scale from baseline to end of intervention at 12 weeks. The scores on the Emotion Reactivity Scale range from 0-84, with a higher score indicating greater emotional reactivity.
Mean change from Baseline in somatization scores on the somatization subscale of Symptom Check-List-90 at 12 weeks | from baseline to end of intervention at 12 weeks
  Changes of somatization scores are measured by the somatization subscale of Symptom Check-List-90 from baseline to end of intervention at 12 weeks. Scores on the somatization subscale of Symptom Check-List-90 range from 0-48, with a higher score indicating greater somatization.

CONTACTS AND LOCATIONS:
Overall Officials: Tatia Lee, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi D, Wong NML, Shao R, Man ISC, Wong CHY, Yuen LP, Chan CCH, Lee TMC. Qigong exercise enhances cognitive functions in the elderly via an interleukin-6-hippocampus pathway: A randomized active-controlled trial. Brain Behav Immun. 2021 Jul;95:381-390. doi: 10.1016/j.bbi.2021.04.011. Epub 2021 Apr 17. PMID 33872709